CLINICAL TRIAL: NCT01895829
Title: Pilot Feasibility Study of Iron Oxide Nanoparticle Magnetic Resonance Dynamic Contrast Enhanced MRI for Primary and Nodal Tumor Imaging in Locally Advanced Head and Neck Squamous Cell Carcinomas
Brief Title: Ferumoxytol - Iron Oxide Nanoparticle Magnetic Resonance Dynamic Contrast Enhanced MRI
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-1127; NCI-2013-02182 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-03; First posted 2013-07-11 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Squamous cell carcinomas of the head and neck; HNSCC; Magnetic resonance imaging; MRI; Ferumoxytol; Ultra-small superparamagnetic iron oxide nanoparticle; USPIO; Contrast agent; Dynamic contrast imaging; DCI
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Magnetic Resonance Spectroscopy; Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ferumoxytol + Magnetic Resonance Imaging (MRI) (Experimental): On Day 1, patient will have 2 standard MRIs, as part of standard of care. About an hour after these 2 scans, patient receives ferumoxytol by vein. Right after that, first study MRI performed. The study MRI performed in the same way that a standard MRI is performed.
  On Day 2, about 24 hours after patient receives ferumoxytol, second study MRI performed.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Drug: Ferumoxytol

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — On Day 1, patient will have 2 standard MRIs, as part of standard of care. About an hour after these 2 scans, patient receives ferumoxytol by vein. Right after that, first study MRI performed. On Day 2, about 24 hours after patient receives ferumoxytol, second study MRI performed.
  Other Names: MRI
Drug: Ferumoxytol — On Day 1, patient will have 2 standard MRIs, as part of standard of care. About an hour after these 2 scans, patient receives ferumoxytol by vein.

SUMMARY:
The goal of this clinical research study is to learn if ferumoxytol, when given at the time of a magnetic resonance imaging (MRI), can help researchers learn more about the spread of certain kinds of cancers.

Ferumoxytol is designed to deliver iron to treat iron-deficiency anemia (low red blood cell counts) in patients with chronic kidney disease. In this study, it will be used as an MRI contrast. Contrasts are used by doctors in order to see MRI images more clearly.

DETAILED DESCRIPTION:
Study Scans:

If you are found to be eligible to take part in this study, you will have 2 study MRIs. These scans will be performed at the Center for Advanced Biomedical Imaging (CABI), in the South Campus Research Building at MD Anderson.

On Day 1, you will have 2 standard MRIs, as part of your standard of care. About an hour after these 2 scans, you will receive ferumoxytol by vein. Right after that, you will have your first study MRI. The study MRI will be performed in the same way that a standard MRI is performed.

On Day 2, about 24 and 72 hours after you receive ferumoxytol, you will have a second study MRI.

Additional Tests:

On Days 1 and 3, as well as 4 weeks after the first study MRI:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests and/or to check your iron level.

On Day 2:

* You will have a physical exam.
* If you have not had one in the last month, you will have a PET-CT scan to check the status of the disease.

Length of Study:

You will be on study for about 4 weeks. You will be taken off study if you have intolerable side effects or you are unable to have the scans for any reason.

This is an investigational study. Ferumoxytol is commercially available and FDA-approved for the treatment of iron deficiency anemia.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older with histologically or cytologically confirmed head and neck squamous cell carcinoma or melanoma
2. Measurable clinical and/or radiographic poly-nodal disease defined as stage N2b, N2c or N3 disease with multiple involved lymph nodes as defined by the American Joint Committee on Cancer (AJCC) cancer staging criteria
3. Patients who have received or are dispositioned to receive a Positron emission tomography (PET) and computerized tomography (CT) [PET-CT] scan within two weeks of starting definitive therapy for their head and neck malignancy and their participation in this study. This implies patients must receive a PET-CT to be eligible for the study.

Exclusion Criteria:

1. Patients who have undergone definitive resection of their primary or nodal disease as well as any chemotherapy or radiation therapy for their head and neck primary tumor.
2. Patients unable or unwilling to give written, informed consent or to undergo MRI imaging.
3. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]). Male partners must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.
4. Patients unable to tolerate DCE-MRI or having an estimated GFR < 60 ml/min/1.73m^2.
5. Contraindications to iron supplementation include hemochromatosis, colitis, history of GI bleeds, alcoholism, or liver disease. Ferumoxytol is contraindicated in patients with evidence of iron overload and/or known hypersensitivity to Feraheme or any of its components. Consequently, we will plan to exclude patients who have symptoms or signs that might be caused by iron overload. These include patients with (unexplained): arthritis (including premature osteoarthritis), congestive heart failure or cardiomyopathy, adult-onset diabetes, secondary hypogonadism, increased skin pigmentation, or patients with persistently elevated serum ferritin not explained by an underlying inflammatory/systemic disease, unless these patients demonstrate a fasting transferrin saturation </= 0.45.
6. Patients with any evidence of iron overload on pre-imaging laboratory studies.
7. Patients with any contraindications to gadolinium-based contrast agents.
8. Patients with claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of Using Ferumoxytol with Magnetic Resonance Imaging (MRI) | 2 days
  Feasibility defined as at least 15 (75%) patients finish the imaging process and good quality images obtained. Good quality image defined as subjective quality assessment score of 4 by two independent radiation oncologists and one radiologist for clinical usability for radiotherapy planning on a 5-point scale. The 5-point scale is defined with 0 implying unable to assess and 5 implying optimal image quality.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Fuller, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org